CLINICAL TRIAL: NCT04843579
Title: A Phase 2, Open-Label, Single-Arm Study of Selinexor in Combination With Clarithromycin, Pomalidomide and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Treatment of Selinexor in Combination With Clarithromycin, Pomalidomide and Dexamethasone for Relapsed Refractory Multiple Myeloma Patients
Acronym: ClaSPd
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-12023093
Record Dates: First submitted 2021-04-10; First posted 2021-04-13 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Myeloma Multiple; Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — selinexor; Clarithromycin; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd) (Experimental): Selinexor
  • Given orally at a dose of 60 mg on days 1, 8, and 15 of a 28-day cycle.
  Dexamethasone
  * Given orally at a dose of 40 mg on days 1, 8, 15 and 22 of a 28-day cycle.
  * Subjects will receive a prescription for dexamethasone 4 mg tablets (generic).
  Clarithromycin
  * Given orally at a dose of 500 mg twice a day on days 1-28 of a 28-day cycle.
  * Subjects will receive a prescription for clarithromycin 250 or 500 mg tablets (generic) for oral administration.
  Pomalidomide
  * Given orally at a dose of 4 mg daily on days 1-21 of a 28-day cycle.
  * Subjects will receive a 21-day supply of pomalidomide 1, 2, 3, or 4 mg capsules for oral administration for each treatment cycle.
  Interventions: Drug: Selinexor; Drug: Clarithromycin; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Given as 60 mg oral capsule
Drug: Clarithromycin — Given as 500 mg oral capsule
Drug: Pomalidomide — Given as 4 mg oral capsule
Drug: Dexamethasone — Given as 40 mg oral capsule

SUMMARY:
The purpose of this study is to determine the efficacy and safety of investigational combination therapy of Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd) for patients with relapsed/refractory multiple myeloma. The hypothesis is that the addition of Selinexor to Clarithromycin, Pomalidomide and Dexamethasone will increase the overall response rate of patients with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines.
* Age ≥18 and <75 years at the time of informed consent.
* Confirmed diagnosis of multiple myeloma
* Symptomatic multiple myeloma per IMWG guidelines.
* Measurable disease as defined by at least one of the following: a. Serum M-protein ≥ 0.5 g/dL by serum protein electrophoresis (SPEP) or, for IgA myeloma, by quantitative IgA, and/or b. Urinary M-protein excretion at least 200 mg/24 hours, and/or c. Serum FLC ≥ 100 mg/L, provided that FLC ratio is abnormal, and/or d. If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement (e.g., for IgA MM), then quantitative Ig levels by nephelometry or turbidimetry are acceptable.
* Relapsed and refractory multiple myeloma with documented evidence of PD after achieving at least SD for ≥ 1 cycle during a previous MM regimen (i.e., relapsed MM), and ≤ 25% response (i.e., patients never achieved ≥ MR) or PD during or within 60 days from the end of the most recent MM regimen (i.e., refractory MM).
* Previously received one to four prior lines of therapy and be pomalidomide-naïve.

Exclusion Criteria:

* Documented active systemic light chain amyloidosis.
* Active plasma cell leukemia.
* Eastern Cooperative Oncology Group (ECOG) Performance Status greater than 2.
* Persistent non-hematological toxicity (except for peripheral neuropathy) from a prior treatment which has not resolved to at least Grade 2 or better by Cycle 1 Day 1 (C1D1).
* Severe hepatic dysfunction with either: a. Total bilirubin > 2x ULN (> 3x ULN in subjects with Gilbert's syndrome [hereditary indirect hyperbilirubinemia]), and/or b. AST and/or ALT > 2.5x ULN
* Severe renal dysfunction with an estimated creatinine clearance of < 15 mL/min calculated using the Cockcroft and Gault formula.
* Impaired hematopoietic function with either: a. White blood cell count < 1,500/mm3, and/or b. Absolute neutrophil count < 1000/mm3, and/or c. Hemoglobin < 8.0 g/dL, and/or d. Platelet count < 100,000/mm3 (for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells, platelets ≥ 75,000/mm3 are acceptable).
* Blood (or blood product) transfusions or blood growth factors within 7 days of C1D1. Use of hematopoietic growth factor support is acceptable, including erythropoietin (EPO), darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), and platelet stimulators (e.g., eltrombopag or romiplostim). However, patients must be platelet transfusion independent for > 1 week in order to be enrolled in the study.
* Radiation, chemotherapy or immunotherapy, or any other anticancer therapy within 2 weeks prior to C1D1, or radio-immunotherapy within 6 weeks prior to C1D1. Patients on long-term glucocorticoids during Screening do not require a washout period. Prior radiation is permitted for treatment of fractures or to prevent fractures, as well as for pain management.
* Patients with history of spinal cord compression with residual paraplegia.
* Treatment with an investigational anti-cancer therapy within 3 weeks prior to C1D1.
* Prior autologous stem cell transplantation < 1 month, or allogeneic stem cell transplantation < 3 months prior to C1D1.
* Active graft versus host disease after allogeneic stem cell transplantation.
* Life expectancy < 3 months.
* Major surgery within 4 weeks prior to C1D1.
* Active, unstable cardiovascular function with either: a. Symptomatic ischemia, b. Uncontrolled clinically significant conduction abnormalities (e.g., patients with ventricular tachycardia on antiarrhythmics are excluded; patients with 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), c. Congestive heart failure (CHF) of New York Heart Association (NYHA) Class ≥ 3, d. Myocardial infarction (MI) within 6 months prior to C1D1, or e. Screening 12-lead ECG showing a baseline QT interval as corrected by Bazett's formula (QTc) > 470 msec
* Uncontrolled active hypertension
* Venous thromboembolism within 6 months prior to C1D1 or a known inherited thrombophilia
* Inability to receive either prophylactic or therapeutic anticoagulation as determined appropriate by the Investigator
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to C1D1
* Any active gastrointestinal dysfunction that prevents the patient from swallowing tablets or interferes with absorption of study treatment
* Currently pregnant or breastfeeding. Lactating females must agree not to breast feed while receiving selinexor, pomalidomide and/or clarithromycin
* A serious psychiatric or medical condition which, in the opinion of the Investigator, could interfere with treatment
* Hypersensitivity or contraindication to selinexor, pomalidomide, dexamethasone and/or clarithromycin
* Prior exposure to a SINE compound, including selinexor
* Concomitant use of any strong CYP3A4 and/or CYP1A2 inhibitors (see Appendix 1)
* Unable to obtain commercial clarithromycin, pomalidomide and dexamethasone through a regular and/or specialty pharmacy.
* Unable or unwilling to register into the mandatory POMALYST REMSTM program and comply with its requirements.
* Male and female patients unwilling or unable to use effective methods of contraception throughout the study and for three months following the last dose. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. Note that female patients of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at Screening and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Monge, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Weill Cornell Medicine - Multiple Myeloma Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd): Selinexor
  • Given orally at a dose of 60 mg on days 1, 8, and 15 of a 28-day cycle.
  Dexamethasone
  * Given orally at a dose of 40 mg on days 1, 8, 15 and 22 of a 28-day cycle.
  * Subjects will receive a prescription for dexamethasone 4 mg tablets (generic).
  Clarithromycin
  * Given orally at a dose of 500 mg twice a day on days 1-28 of a 28-day cycle.
  * Subjects will receive a prescription for clarithromycin 250 or 500 mg tablets (generic) for oral administration.
  Pomalidomide
  * Given orally at a dose of 4 mg daily on days 1-21 of a 28-day cycle.
  * Subjects will receive a 21-day supply of pomalidomide 1, 2, 3, or 4 mg capsules for oral administration for each treatment cycle.
  Selinexor: Given as 60 mg oral capsule
  Clarithromycin: Given as 500 mg oral capsule
  Pomalidomide: Given as 4 mg oral capsule
  Dexamethasone: Given as 40 mg oral capsule
Period: Overall Study
Arm/Group | Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd)
Started | 4
Completed | 2
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response Rate of Partial Response or Better
Description: ORR is defined as participants who experience a partial response, very good partial response, complete response, or stringent complete response per International Myeloma Working Group Criteria (IMWG) 2016 criteria. Complete Response is defined as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. Stringent Complete Response is defined as complete response as noted previously plus normal free light chain ratio and absence of clonal cells in bone marrow biopsy by immune-histochemistry. Partial Response is ≥50% reduction of serum M-protein plus reduction in 24 hour urinary M-protein by ≥90% or to <200 mg per 24 h. Very Good Partial Response is serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hr.
Time Frame: Until disease progression; the maximum time any participant was followed for ORR was 287 days
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd)
Number analyzed (Participants) | 4
Participants | 2

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be determined by Events as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The frequency of adverse events will be collected in tabular summary from when a participant consent to study until end of study or patient participant starts a new treatment.
Time Frame: Adverse events were collected from time of informed consent until 30 days after the last day of study drug administration for each participant. The maximum period that AEs were collected for a participant was 300 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd)
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of informed consent until 30 days after the last day of study drug administration for each participant. The maximum period that AEs were collected for a participant was 300 days.
Arm/Group | Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd) (N=4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor, Clarithromycin, Pomalidomide and Dexamethasone (ClaSPd) (N=4)
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Blurred vision (Eye disorders) | 1
Concentration Impairment (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
COVID-19 Infection (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Gait Disturbance (General disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Lymphocyte Count Decreased (Investigations) | 1
Mucosal Infection (Infections and infestations) | 1 — Oral thrush
Nausea (Gastrointestinal disorders) | 1
Neutrophil Count Decreased (Investigations) | 2
Platelet Count Decreased (Investigations) | 2
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 — Achilles tendon pain
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Mania (Renal and urinary disorders) | 1 — Steroid-related
Upper Respiratory Infection (Infections and infestations) | 1
Weight Gain (Investigations) | 1

LIMITATIONS AND CAVEATS:
The statistical analysis plan (and associated statistical power) was based on an expected sample size of 26 participants. As only 4 participants enrolled, this reduced sample size was not sufficient for the statistical analysis plan as written, and, therefore, only descriptive statistics for the response proportions can be presented for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT04843579/Prot_SAP_000.pdf